CLINICAL TRIAL: NCT00753922
Title: Core Gel Study of the Safety and Effectiveness of Mentor Round Low Bleed Silicone Gel-filled Mammary Prostheses in Patients Who Are Undergoing Primary Breast Augmentation, Primary Breast Reconstruction or Revision
Brief Title: Core Gel Study of the Safety and Effectiveness of Mentor Round Low Bleed Silicone Gel-filled Mammary Prostheses
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mentor Worldwide, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-009-0799-01
Expanded Access: NCT00948948 (Approved for marketing)
Record Dates: First submitted 2008-09-15; First posted 2008-09-17 (Estimated); Results first posted 2013-08-23 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-03

CONDITIONS: Breast Reconstruction; Breast Augmentation; Breast Revision
Keywords: Breast Reconstruction; Breast Augmentation; Revision; Silicone breast implants; Round low-bleed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Primary Augmentation (Other): The Augmentation cohort will include patients who have post-lactational mammary involution or wish general breast enlargement.
  Interventions: Device: Mentor Round Low Bleed Gel-filled Mammary Protheses, both Siltex and Smooth Surface
- Primary Reconstruction (Other): The Reconstruction cohort will include patients with loss of breast due to mastectomy or with deformities secondary to disease, malignancy, trauma, and congenital deformity.
  Congenital deformities will include deformities of the breast itself as well as skeletal abnormalities reflected in breast deformity or asymmetry.
  Interventions: Device: Mentor Round Low Bleed Gel-filled Mammary Protheses, both Siltex and Smooth Surface
- Revison Augmentation (Other): Patients in this cohort will have had previous breast augmentation with silicone or saline filled implants and are having a revision surgery to correct or improve the result of any previous breast augmentation surgery.
  Interventions: Device: Mentor Round Low Bleed Gel-filled Mammary Protheses, both Siltex and Smooth Surface
- Revision Reconstruction (Other): Patients in this cohort will have had previous breast reconstruction with silicone or saline filled implants and are having a revision surgery to correct or improve the result of any previous breast reconstruction surgery.
  Interventions: Device: Mentor Round Low Bleed Gel-filled Mammary Protheses, both Siltex and Smooth Surface

INTERVENTIONS:
Device: Mentor Round Low Bleed Gel-filled Mammary Protheses, both Siltex and Smooth Surface — Two types of Mentor Round Low-Bleed Silicone Gel-filled Mammary Prostheses will be used in the study: the Siltex textured surface device and the smooth surface device. Each implant is a silicone elastomer (rubber) mammary device that is supplied individually packaged in a doubled wrapped packaging system, sterile, and non-pyrogenic (does not cause fever). Each device consists of a silicone shell encasing a silicone gel filler material with a patch on the posterior side of the device. The basic smooth device shell consists of a silicone layer sandwiched in between two other silicone layers. This construction acts as a barrier to slow the diffusion of (spread) any gel filler materials through the shell. The Siltex textured shell consists of a smooth shell to which is bonded an additional layer of silicone with a textured pattern imprinted into its surface. The Siltex shell is intended to prevent tissue ingrowth. The implants will be available in sizes 100cc through 800ccs.

SUMMARY:
The Core Gel Study is designed to demonstrate safety and effectiveness of Mentor's Round Low-Bleed Silicone Gel-filled Mammary Prostheses in women who are undergoing primary augmentation, primary reconstruction, or revision. Safety information on the rate of capsular contracture, rupture, and infection will be collected, and used to help determine device safety.

Approximately 1000 patients at centers across the United States will be enrolled in this research study. These patients will be implanted with silicone breast prostheses and monitored for 10 years to collect information on risks associated with the implant surgery as well as changes in the way these patients feel about themselves.

DETAILED DESCRIPTION:
Silicone gel-filled breast implants were introduced in the early sixties and were in wide-scale distribution by the time the Medical Device Amendments to the Food Drug and Cosmetic Act was passed in 1976. In 1983, gel-filled breast implants were designated as Class III devices requiring premarket approval. In May 1990, the Food and Drug Administration (FDA) published a proposed request (515(b)) for Premarket Approval Applications (PMA) and in April 1991 published the final request. This final publication put manufacturers of gel-filled breast implants on notice that for continued marketing of gel-filled breast implants, a PMA was due to FDA in 90 days from the final publication date.

A premarket approval (PMA) for the Mentor gel-filled breast implants was filed with the FDA in July 1991. At the FDA General and Plastic Surgery Advisory Committee meeting in November 1991, the committee recommended the submission of additional information to establish the safety and effectiveness of gel-filled breast implants.

In January 1992, the FDA Commissioner announced a voluntary moratorium of the sale of gel-filled breast implants to allow the advisory panel time to assess additional information. In April 1992, the moratorium was lifted but only for reconstruction and revision patients. Every patient implanted had to be part of an adjunct study, and had to be offered participation in a registry of gel-filled breast implant patients. In order to be implanted with gel-filled implants for augmentation, women had to be enrolled in a core clinical study.

The objective of this study is to determine the safety and effectiveness of the smooth and textured surface Mentor Round Low-Bleed Silicone Gel-filled Mammary Prostheses in women who are undergoing primary breast augmentation, primary breast reconstruction or revision.

ELIGIBILITY:
Inclusion Criteria:

* Subject is Genetic female and at least 18 years old
* A candidate for:
* Primary breast augmentation (for post-lactational mammary involution or general breast enlargement)
* Primary breast reconstruction (for cancer, trauma, surgical loss of breast or congenital deformity)
* Revision surgery (previous augmentation or reconstruction with silicone-filled or saline-filled implants)
* Signs the Informed Consent
* Agrees to follow the procedures for explant analysis
* Agrees to comply with follow-up procedures, including returning for all follow-up visits

Exclusion Criteria:

* Patient is pregnant
* Has nursed a child within three months of study enrollment
* Been implanted with any silicone implant other than breast implants (e.g. silicone artificial joints or facial implants)
* Confirmed diagnosis of the following rheumatic diseases or syndromes: SLE, Sjogren's syndrome, scleroderma, polymyositis, or any connective tissue disorder, rheumatoid arthritis, crystalline arthritis, infections arthritis, spondylarthropathies, any other inflammatory arthritis, osteoarthritis, fibromyalgia, or chronic fatigue syndrome
* Currently has a condition that could compromise or complicate wound healing (except reconstruction patients)
* Patient in Augmentation cohort and has diagnosis of active cancer of any type
* Infection or abscess anywhere in the body
* Demonstrates tissue characteristics which are clinically incompatible with implant (e.g. tissue damage resulting from radiation, inadequate tissue, or compromised vascularity)
* Possesses any condition, or is under treatment for any condition which, in the opinion of the investigator and/or consulting physicians(s), may constitute an unwarranted surgical risk
* Anatomic or physiologic abnormality which could lead to significant postoperative adverse events
* Demonstrates characteristics that are unrealistic/unreasonable with the risks involved with the surgical procedure
* Premalignant breast disease without a subcutaneous mastectomy
* Untreated or inappropriately treated breast malignancy, without mastectomy
* Implanted metal or metal devices, history of claustrophobia or other condition that would make a MRI scan prohibitive

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1008 (Actual)
Dates: Start 2000-09; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Mentor Worldwide, LLC, Santa Barbara, California, United States

REFERENCES:
- [Derived] Caplin DA, Calobrace MB, Wixtrom RN, Estes MM, Canady JW. MemoryGel Breast Implants: Final Safety and Efficacy Results after 10 Years of Follow-Up. Plast Reconstr Surg. 2021 Mar 1;147(3):556-566. doi: 10.1097/PRS.0000000000007635. PMID 33620918
- [Derived] Caplin DA. Indications for the use of MemoryShape breast implants in aesthetic and reconstructive breast surgery: long-term clinical outcomes of shaped versus round silicone breast implants. Plast Reconstr Surg. 2014 Sep;134(3 Suppl):27S-37S. doi: 10.1097/PRS.0000000000000609. PMID 25158767

RESULTS

PARTICIPANT FLOW:
Groups:
- Primary Reconstruction: The Reconstruction cohort will include patients with loss of breast due to mastectomy or with deformities secondary to disease, malignancy, trauma, and congenital deformity.
  Congenital deformities will include deformities of the breast itself as well as skeletal abnormalities reflected in breast deformity or asymmetry.
  Asymmetry is one or more of the following conditions:
  * One cup size difference in breast size.
  * The need to differentially pad one bra cup to match the opposite breast size.
  * Asymmetry due to chest wall deformity such as scoliosis or other deformities of the thoracic cage and/or associated visible differences in shoulder height that can make one breast appear to be at a different height than the other.
- Revision Augmentation: Patients in this cohort will have had previous breast augmentation or reconstruction with silicone or saline filled implants.
Period: Overall Study
Arm/Group | Primary Augmentation | Primary Reconstruction | Revision Augmentation | Revision Reconstruction
Started | 552 | 251 | 145 | 60
Completed | 306 | 157 | 82 | 37
Not Completed | 246 | 94 | 63 | 23
Not completed — Lost to Follow-up | 155 | 24 | 28 | 5
Not completed — Withdrawal by Subject | 9 | 11 | 4 | 2
Not completed — Patient Non-compliance | 55 | 22 | 14 | 11
Not completed — Patients Not Completing Visit | 11 | 0 | 1 | 0
Not completed — Death | 2 | 23 | 2 | 1
Not completed — Discontinuation Due to Explantation | 14 | 14 | 14 | 4

BASELINE CHARACTERISTICS:
Population: All enrolled subjects are included
Groups:
- Total: Total of all reporting groups
Arm/Group | Primary Augmentation | Primary Reconstruction | Revision Augmentation | Revision Reconstruction | Total
Number analyzed (Participants) | 552 | 251 | 145 | 60 | 1008
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 551 | 245 | 145 | 54 | 995
  >=65 years | 1 | 6 | 0 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.5 (8.09) | 45.3 (10.87) | 41.8 (9.66) | 50.8 (10.82) | 39.2 (10.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 552 | 251 | 145 | 60 | 1008
  Male | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 552 | 251 | 145 | 60 | 1008

OUTCOME MEASURES:

1. Primary Outcome: 10-Year Kaplan-Meier Estimated Cumulative Incidence Rate of Occurrence of Any Reoperation
Description: Time of occurrence calculated as the number of days from the date of the implant procedure to the onset date of the event. Patients were censored as of the date of their last office visit, the 120 month time point, or the date of explantation of all initial study devices, whichever was earliest.
Time Frame: 10 years
Population: All enrolled subjects are included
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Groups:
- Revison Augmentation: Patients in this cohort will have had previous breast augmentation or reconstruction with silicone or saline filled implants.
Arm/Group | Primary Augmentation | Primary Reconstruction | Revison Augmentation | Revision Reconstruction
Number analyzed (Participants) | 552 | 251 | 145 | 60
percentage of subjects | 25.5 [21.9 to 29.5] | 49.0 [42.6 to 55.7] | 43.6 [35.8 to 52.4] | 50.7 [38.7 to 64.0]

2. Primary Outcome: Overall Mean Change in Circumferential Chest Size
Description: Change in Chest Size was calculated by subtracting the chest circumference prior to surgery from the chest circumference measured at the end of the study
Time Frame: Change from baseline to 10 years post-baseline
Population: All enrolled subjects
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Primary Augmentation | Primary Reconstruction | Revison Augmentation | Revision Reconstruction
Number analyzed (Participants) | 552 | 251 | 145 | 60
centimeters | 7.45 (4.50) | 4.88 (7.25) | 2.89 (4.56) | 4.18 (5.68)

3. Primary Outcome: 10-Year Kaplan-Meier Estimated Cumulative Incidence Rate of Occurrence of Baker III, IV Capsular Contracture
Description: Baker III was identified as "firm with visible distortion" and Baker IV was identified as "obvious spherical distortion". Time of occurrence calculated as the number of days from the date of the implant procedure to the onset date of the event. Patients were censored as of the date of their last office visit, the 120 month time point, or the date of explantation of all initial study devices, whichever was earliest.
Time Frame: 10 Years
Population: All enrolled subjects
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Primary Augmentation | Primary Reconstruction | Revison Augmentation | Revision Reconstruction
Number analyzed (Participants) | 552 | 251 | 145 | 60
percentage of subjects | 12.1 [9.6 to 15.2] | 20.5 [15.5 to 26.7] | 24.4 [18.1 to 32.5] | 36.9 [25.0 to 52.2]

4. Primary Outcome: 10-Year Kaplan-Meier Estimated Cumulative Incidence Rate of Occurrence of Infection
Description: as for outcome 1
Time Frame: 10 Years
Population: All enrolled subjects
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Primary Augmentation | Primary Reconstruction | Revison Augmentation | Revision Reconstruction
Number analyzed (Participants) | 552 | 251 | 145 | 60
percentage of subjects | 1.6 [0.9 to 3.1] | 6.2 [3.8 to 10.1] | 1.4 [0.4 to 5.5] | 0.0 [NA to NA] — Since there were no Infections observed in this arm, the 95% Confidence is not estimable under the Kaplan-Meier framework.

5. Primary Outcome: 10-Year Kaplan-Meier Estimated Cumulative Incidence Rate of Occurrence of Explantation With or Without Replacement
Description: as for outcome 1
Time Frame: 10 Years
Population: All enrolled subjects
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Primary Augmentation | Primary Reconstruction | Revison Augmentation | Revision Reconstruction
Number analyzed (Participants) | 552 | 251 | 145 | 60
percentage of subjects | 11.6 [9.1 to 14.8] | 33.4 [27.6 to 40.1] | 24.1 [17.7 to 32.3] | 37.8 [26.7 to 51.7]

6. Post Hoc Outcome: 10-Year Kaplan-Meier Estimated Cumulative Incidence Rate of Occurrence of Complications
Description: The safety analyses were conducted in accordance with the FDA November 17, 2006 "Guidance for Industry and FDA Staff - Saline, Silicone Gel, and Alternative Breast Implants." The study investigator assessed any complications durign study follow-up visits in alignment with this guidance. Time of occurrence was calculated as the number of days from the date of the implant procedure to the onset date of the event. Patients were censored as of the date of their last office visit, the 120 month time point, or the date of explantation of all initial study devices, whichever was earliest. Complications with an incidence > 5.0% are reported.
Time Frame: 10 years
Population: All Enrolled Subjects
Measure: Number (95% Confidence Interval); unit: percentage of subjects
Arm/Group | Primary Augmentation | Primary Reconstruction | Revison Augmentation | Revision Reconstruction
Number analyzed (Participants) | 552 | 251 | 145 | 60
percentage of subjects
  Breast Mass | 5.6 [3.9 to 7.9] | 8.6 [5.5 to 13.4] | 6.0 [3.0 to 11.6] | 5.1 [1.7 to 15.1]
  Breast Pain | 2.9 [1.8 to 4.8] | 5.2 [2.9 to 9.2] | 3.2 [1.2 to 8.2] | 5.2 [1.7 to 15.2]
  Metastatic Disease | 0 [0 to 0] | 6.9 [4.2 to 11.2] | 0 [0 to 0] | 3.8 [1.0 to 14.6]
  Nipple Sensation Changes | 12.8 [10.2 to 16.0] | 2.1 [0.9 to 5.0] | 13.6 [8.9 to 20.4] | 4.0 [1.0 to 15.2]
  Implant Malposition/Displacement | 1.0 [0.4 to 2.5] | 2.3 [1.0 to 5.5] | 2.3 [0.7 to 7.0] | 6.7 [2.6 to 16.9]
  Lack of Projection | 0 [0 to 0] | 1.0 [0.3 to 4.2] | 0 [0 to 0] | 5.5 [1.8 to 16.3]
  Patient Dissatisfaction | 0.4 [0.1 to 1.5] | 4.8 [2.5 to 9.2] | 3.6 [1.5 to 8.5] | 9.0 [3.4 to 23.0]

ADVERSE EVENTS:
Time Frame: Baseline to 10 Years.
Description: Adverse events were not coded according to the MedDRA dictionary, rather they were collected as Complications in alignment with the 2006 FDA Guidance. Safety endpoints are summarized under Primary, Secondary, and Post-Hoc Outcome Measures. All complications with a frequency above 5% are reported in the Outcome Measures section.
Arm/Group | Primary Augmentation | Primary Reconstruction | Revison Augmentation | Revision Reconstruction
Serious Adverse Events (participants affected / at risk) | 0/552 | 0/251 | 0/145 | 0/60
Other Adverse Events (participants affected / at risk) | 0/552 | 0/251 | 0/145 | 0/60

LIMITATIONS AND CAVEATS:
Adverse events were not coded according to the MedDRA dictionary, rather they were collected as Complications in alignment with the 2006 FDA Guidance for Industry and FDA Staff - Saline, Silicone Gel, and Alternative Breast Implants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor acknowledges that the Investigator and his/her collaborators shall be free to publish the background, methods and results of their own research without restraint. Prior review of any proposed manuscript or abstract will be provided to Sponsor to prevent premature disclosure of trade secrets or proprietary information. The Investigator acknowledges that the Sponsor reserves the right to publish and present the overall study results, including assigning authorship.